CLINICAL TRIAL: NCT06758791
Title: Relationship of Respiratory Muscle Functions With Balance and Gait in Chronic Ischemic Stroke Patients
Brief Title: Respiratory Muscle Functions With Balance and Gait in Stroke Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: University of Beykent (Other)
Responsible Party: Principal Investigator, Sümeyye Akçay, Investigator, Saglik Bilimleri Universitesi
Other Study IDs: BeykentUniversity
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Chronic Stroke; Respiratory Muscles
Keywords: Chronic Stroke; Ischemic; Respiratory Muscles; Pulmonary Funtion Test; Balance; Gait
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke, which can occur due to many different causes and is one of the most common neurological conditions, is one of the main causes of disability worldwide. The most common disorders that occur after stroke are motor disorders. In addition, respiratory problems such as changes in breathing patterns and decreased ventilation function may accompany these patients. Respiratory problems are an important risk factor in the development of long-term mortality for both cardiovascular diseases and stroke. With all these changes, a serious decrease in patients' activity performance is observed. While the focus is on motor function losses in stroke rehabilitation, problems in pulmonary functions do not receive the necessary attention. In stroke rehabilitation, evaluating and treating patients from every perspective will further increase the effectiveness of the treatments applied.

DETAILED DESCRIPTION:
According to WHO, stroke, also known as cerebrovascular accident, is a neurological condition that results in rapidly developing loss of brain function as a result of a problem in the blood supply to the brain. Stroke, which ranks third among the causes of death, is one of the leading causes of disability. Brain damage following stroke affects the central control of respiration, leading to various respiratory disorders. Dysfunction of the main respiratory muscle, the diaphragm, and particularly of the respiratory muscles on the paretic side of the body, is the most common and serious problem, causing asymmetric chest wall movements, changes in respiratory patterns, decreased lung volumes, and pulmonary complications. These changes in respiration cause further decreases in aerobic capacity, walking function, and the ability to perform daily living activities, especially in stroke patients who require an intensive rehabilitation program, and may increase the risk of pulmonary complications. At the same time, this situation may increase the risk of mortality by 2-6 times in stroke patients in the acute phase, prolong the average hospital stay, and worsen neurological dysfunctions. Therefore, evaluation of pulmonary functions and respiratory muscles before rehabilitation is very important to protect patients from possible accompanying pulmonary complications and to increase the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Having had a stroke for the first time
2. Being 18 years of age or older
3. Having an ischemic type of stroke
4. Having had a stroke for at least 6 months
5. Having a Modified Rankin Score of ≥3
6. Being able to communicate
7. Agreeing to participate in the study

Exclusion Criteria:

1. Hemispatial neglect
2. Having a psychiatric disease
3. Having any respiratory problems before the stroke
4. Having any orthopedic, neurological, cardiopulmonary disease that would constitute a contraindication for the protocols to be applied

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic Stroke Patients
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-03-02 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
Respiratory Function Tests | 1 day (It will be performed one time.)
  These are tests used in combination with the clinic to evaluate and grade damage and abnormalities in respiratory system functions. Spirometric measurement reflects the time, volume and flow values measured during normal breathing, forced inspiration, forced expiration, deep and rapid breathing for a certain period of time. The test is evaluated by comparing the basal values obtained by creating gender, height, weight and age groups in healthy people in the community where the measurement is made. Lung functions physiologically consist of four volumes. Expiratory reserve volume (ERV), inspiratory reserve volume (IRV), residual volume (RV) and tidal volume (VT). The sum of the four volumes gives the total lung capacity (TLC).

SECONDARY OUTCOMES:
6-Minute Walk Test | 1 day (It will be performed one time.)
  The 6MWT is defined as a submaximal test that can be easily applied to healthy or sick individuals, and is evaluated as an indicator of exercise capacity and walking capacity, as well as many cardiovascular diseases. The 6MWT is referred to as the "Gold Standard" test of walking capacity.
Berg Balance Scale | 1 day (It will be performed one time.)
  A scale consisting of 14 tests that measure the ability to maintain balance during different positions, postural changes and movement. The assessment is based on the person's ability to perform each test independently and/or for a certain time or distance. The rating is made between 0 and 4 points (0: cannot perform, 4: normal performance). The total score varies between 0 (dependent) and 56 (independent).

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Halil Ural, M.D., Principal Investigator — Beykent University; Dudu Kübra Akyol, PT, Study Chair — IAU Medical Park Florya Hospital; Sümeyye Akçay, PT, Study Chair — Saglik Bilimleri University
Locations (1):
- Beykent Üniversity, Istanbul, Büyükçekmece, Turkey (Türkiye)